CLINICAL TRIAL: NCT00703391
Title: A 2-week, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Tolerability and Pharmacokinetics of Orally Administered AZD9668 in Patients With COPD
Brief Title: A Two Week Study to Assess the Tolerability of AZD9668 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0520C00002
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2010-12-29 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic; obstructive; pulmonary; lung; respiratory disease; tolerability; placebo-controlled; pharmacokinetics; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Respiration Disorders | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active Treatment
  Interventions: Drug: AZD9668
- 2 (Placebo Comparator): Placebo Treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9668 — 30mg oral tablets twice daily (bid) for 14 days
  Arms: 1
Drug: Placebo — Matched placebo to 30mg oral tablet twice daily (bid) for 14 days
  Arms: 2

SUMMARY:
The purpose of this study is to assess the tolerability (effect of drug on body) and pharmacokinetics (effect of body on drug) of AZD9668 in patients with mild to moderate COPD

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate COPD
* Smokers or ex-smokers
* post-menopausal females

Exclusion Criteria:

* Past history or current evidence of clinically significant heart disease
* Lung disease other than COPD
* Treatment with systemic steroids within 8 weeks of study visit 2
* Treatment with antibiotics within 4 weeks of study visit 1 or study visit 2

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Panke, Principal Investigator — Parexel International GmbhH (CRO)
Locations (1):
- Research Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 11 June 2008. Last patient completed: 09 October 2008. Single-centre study performed at a Clinical Pharmacology Unit
Groups:
- AZD9668: AZD9668 2x30mg oral tablets twice daily (bid) for 14 days
- Placebo: Matched placebo tablets twice daily (bid) for 14 days
Period: Overall Study
Arm/Group | AZD9668 | Placebo
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9668 | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age Continuous [Mean (Full Range); unit: Years] | 57.6 [42 to 70] | 52.8 [44 to 65] | 56 [42 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Alanine Aminotransferase (ALT)
Description: ALT level greater than 3 times the upper limit of normal
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 0 | 0

2. Primary Outcome: Aspartate Aminotransferase (AST)
Description: AST level greater than 3 times the upper limit of normal
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 0 | 0

3. Primary Outcome: Creatine Kinase (CK)
Description: Change from baseline to Day 14
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
IU/L | 2.57 (19.260) | -69.57 (141.383)

4. Primary Outcome: Total Bilirubin
Description: Change from baseline to Day 14
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
micromol/L | 0.11 (2.124) | -0.28 (2.563)

5. Primary Outcome: Creatinine
Description: Creatinine level greater than the upper limit of normal
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 1 | 1

6. Primary Outcome: Haemoglobin (Hb)
Description: Change from baseline to Day 14
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
g/L | -2.0 (4.73) | -0.2 (6.18)

7. Primary Outcome: Reticulocytes
Description: Change from baseline to Day 14
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Mean (Standard Deviation); unit: relative particle count (%)
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
relative particle count (%) | -0.15 (2.851) | 1.73 (1.605)

8. Primary Outcome: Leucocytes
Description: Change from baseline to Day 14
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Mean (Standard Deviation); unit: 10**9/L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
10**9/L | -0.001 (0.8816) | 0.265 (0.4657)

9. Primary Outcome: QTcF (QT Interval Corrected for Heart Rate by Fridericia's Method)
Description: QTcF interval greater than 450 ms
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 0 | 0

10. Primary Outcome: QTcF
Description: QTcF change from baseline greater than 60 ms
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 0 | 0

11. Secondary Outcome: Sputum Absolute Neutrophil Count
Description: Change from baseline to Day 14 in absolute neutrophil count
Time Frame: Pre-dose day -1 to post-dose on day 14
Measure: Median (Full Range); unit: 10**9/L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 7 | 4
10**9/L | -0.4890 [-1.439 to 0.439] | -2.5645 [-9.198 to -0.283]

12. Secondary Outcome: Sputum Differential Neutrophil Count
Description: Change from baseline to Day 14 in percentage neutrophil count
Time Frame: Pre-dose day -1 to post-dose on day 14
Measure: Median (Full Range); unit: Percentage
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Percentage | 1.8 [-11.0 to 10.0] | -4.25 [-9.0 to 8.7]

13. Secondary Outcome: AZD9668 Sputum Concentrations
Time Frame: Pre-dose day -1 to post-dose on day 14
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 11 | 0
nM | 41.7 [26.5 to 64.3] |

14. Secondary Outcome: Quantitative Sputum Bacteriology
Description: Number of patients with an increase in bacteriological count from Day -1 to Day 15
Time Frame: Pre-dose day -1 to post-dose on day 15
Measure: Number; unit: Participants
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 3 | 2

15. Primary Outcome: FEV1 (Forced Expiratory Volume in the First Second)
Description: Change from baseline to Day 14
Time Frame: Throughout the duration of the study (pre-dose, cmax, steady state, end of dosing and post dose)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 6
L | 0.039 (0.2173) | -0.110 (0.3043)

16. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post-dose (AUC(0-12))
Description: AUC(0-12) following 14 days' dosing
Time Frame: Pre-dose on day -1 to day 15 (end of dosing)
Measure: Geometric Mean (Full Range); unit: nM.h
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 0
nM.h | 7560 [5820 to 9570] |

17. Primary Outcome: Observed Peak or Maximum Plasma Concentration Following Drug Administration (Cmax)
Description: Cmax following 14 days' dosing
Time Frame: Pre-dose on day -1 to day 15 (end of dosing)
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 0
nM | 1420 [1030 to 1930] |

18. Primary Outcome: Time to Reach Observed Peak or Maximum Concentration Following Oral Drug Administration (Tmax)
Description: tmax following 14 days' dosing
Time Frame: Pre-dose on day -1 to day 15 (end of dosing)
Measure: Median (Full Range); unit: hours
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 0
hours | 1.01 [0.490 to 2.01] |

19. Primary Outcome: Terminal Half-life of Drug in Plasma (t1/2)
Description: t1/2 following 14 days' dosing
Time Frame: Pre-dose on day -1 to day 15 (end of dosing)
Measure: Median (Full Range); unit: hours
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 0
hours | 5.89 [5.00 to 6.46] |

20. Primary Outcome: Renal Clearance of Drug From Plasma (CLR)
Description: CLR following 14 days' dosing
Time Frame: Pre-dose on day -1 to day 15 (end of dosing)
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 12 | 0
L/h | 6.13 [3.49 to 8.22] |

ADVERSE EVENTS:
Arm/Group | AZD9668 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 5 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD9668 | Placebo
Palpitations (Cardiac disorders) | 1/12 | 0/6
Diarrhoea (Gastrointestinal disorders) | 1/12 | 0/6
Dyspepsia (Gastrointestinal disorders) | 0/12 | 1/6
Nausea (Gastrointestinal disorders) | 1/12 | 0/6
Vomiting (Gastrointestinal disorders) | 1/12 | 0/6
Chest discomfort (General disorders) | 1/12 | 0/6
Fatigue (General disorders) | 0/12 | 1/6
Respiratory tract infection (Infections and infestations) | 1/12 | 0/6
Back pain (Ear and labyrinth disorders) | 2/12 | 0/6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/12 | 0/6
Headache (Nervous system disorders) | 1/12 | 4/6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/12 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No